CLINICAL TRIAL: NCT01133613
Title: Double-Blind, Randomized, Single Dose Escalation Safety Study of Intraarticular Bone Morphogenic Protein (38A BMP-7) in Subjects With Osteoarthritis (OA) of the Knee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stryker Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 09-OA-003
Record Dates: First submitted 2010-05-27; First posted 2010-05-31 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Bone Morphogenetic Protein 7

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Cohort 1 (Experimental): 0.03 mg/ml BMP-7 or placebo via intraarticular knee injection
  Interventions: Drug: Bone morphogenetic protein 7
- Cohort 2 (Experimental): 0.1 mg/ml BMP-7 or placebo via intraarticular knee injection
  Interventions: Drug: Bone morphogenetic protein 7
- Cohort 3 (Experimental): 0.3 mg/ml BMP-7 or placebo via intraarticular knee injection
  Interventions: Drug: Bone morphogenetic protein 7

INTERVENTIONS:
Drug: Bone morphogenetic protein 7 — Single intraarticular injection of BMP-7 or placebo on Day 1

SUMMARY:
The objective of the study is to determine the safety and tolerability of two different formulations of BMP-7 for the treatment of osteoarthritis of the knee.

ELIGIBILITY:
Inclusion Criteria

* Ambulatory with a diagnosis of OA of the knee with symptoms for at least 6 months and pain on the majority of days in the last 30 days.
* >40 years
* Radiographic evidence of at least one osteophyte in either knee at screening

Exclusion Criteria

* Concurrent medical or arthritis condition that could interfere with evaluation of index knee joint (including fibromyalgia)
* Unwilling to abstain from NSAIDs and/or other analgesic medications for 48 hrs prior to assessments. Subjects can remain on acetaminophen up to 3.0 g daily.
* Received arthroscopic or open surgery to the index knee within 6 months of screening
* History of joint replacement surgery (index knee).
* Corticosteroid, short acting hyaluronic acid, or other intraarticular injections of the index knee within 3 months of screening
* Long acting hyaluronic acid injection of the index knee within 6 months of screening
* History of Reiter's syndrome, rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, lymphoma, and arthritis associated with inflammatory bowel disease, sarcoidosis, amyloidosis or fibromyalgia.
* History of malignancy with the exception of resected basal cell, squamous cell of the skin, resected cervical atypia or carcinoma in situ.
* Female subject with reproductive capability.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-05; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Safety (physical examination, vital signs, clinical laboratory measurements, adverse events) | Baseline, Day 2, Week 1, Week 2, Week 4, Week 8, Week 12, Week 24

SECONDARY OUTCOMES:
WOMAC pain and function | Baseline, Week 4, Week 8, Week 12, Week 24
Patient and physician global VAS | Baseline, Week 1, Week 2, Week 4, Week 8, Week 12, Week 24
Quality of life measurement (SF-36) and pain medication use | Baseline, Week 4, Week 8, Week 12, Week 24

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida Medical Research Institute, Gainesville, Florida
  - Tufts Medical Center, Boston, Massachusetts